CLINICAL TRIAL: NCT04206527
Title: Strengthening People-centered Accessibility, Respect, and Quality for Family Planning Services in India
Brief Title: Improving Person-Centered Care for Family Planning in India
Acronym: SPARQ_FPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Population Services International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-25950
Record Dates: First submitted 2019-12-17; First posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Family Planning
Keywords: Person-Centered Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention - Women (Experimental): Women who receive enhanced FP counseling from an ASHA
  Interventions: Behavioral: Training of AHSAs on PCC for FP
- Control - Women (No Intervention): Women who receive standard FP counseling from an ASHA
- Intervention - ASHA (Experimental): ASHA who receive enhanced FP counseling training
  Interventions: Behavioral: Enhanced FP training
- Control ASHA (No Intervention): ASHA who receive standard FP training

INTERVENTIONS:
Behavioral: Training of AHSAs on PCC for FP — ASHAs provided with training on FP methods and counseling plus PCC for FP
  Arms: Intervention - Women
Behavioral: Enhanced FP training — Participation in an enhanced FP training including PCC
  Arms: Intervention - ASHA

SUMMARY:
To evaluate the impact of a training to ASHAs on person-centered care (PCC) for family planning (FP).

DETAILED DESCRIPTION:
ASHAs will be provided with a training on family planning (FP) counseling and method options. Half of the group will receive additional trainings on person-centered care (PCC) principles and respectful care while the other half of the group will not receive this additional training. Women working with both the control ASHAs (FP trained) and Interventions ASHAs (FP+PCC trained) will be surveyed following their interactions with the ASHA to understand the quality of their experience with the ASHA and whether the woman has taken up a FP method of her choice following interaction with the ASHA.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-49
* Consented/agreed to participate
* Has met with a control or intervention ASHA at least once in the previous three months

Exclusion Criteria:

* Not a women aged 18-49
* Did not consent/agree to participate
* Has not met with a control or intervention ASHA at least once in the previous three months

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1104 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Person-centered Family Planning Scale Score | 3-months after first FP counseling with ASHA
  Survey conducted with women: self-report of experiences of care. Possible range 0-43; higher the score the better the experience of care
Experience of providing FP counseling | at least 3-months after FP training
  In-depth interviews with ASHAs from intervention and control arms to understand experience providing FP counseling

SECONDARY OUTCOMES:
Uptake of Family Planning | 3-months after first FP counseling with ASHA
  Self-report of uptake of a FP method; Yes/No/I Don't remember

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Diamond-Smith, PhD, Study Director — University of California, San Francisco
Locations (1):
- Population Services International, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diamond-Smith N, McDonell C, Sahu AB, Roy KP, Giessler K. A mixed-methods evaluation of the impact of a person-centered family planning intervention for community health workers on family planning outcomes in India. BMC Health Serv Res. 2020 Dec 11;20(1):1139. doi: 10.1186/s12913-020-05995-9. PMID 33308230